CLINICAL TRIAL: NCT06971081
Title: Blue-violet Light Emitting Diode Application Following Dental Extraction in Patients Taking Direct Oral Anticoagulants. A Randomised Controlled Clinical Trial
Brief Title: LED Application Following Dental Extraction in Patients Taking Direct Oral Anticoagulants.
Acronym: DENT-DOAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23/SC/0050
Record Dates: First submitted 2025-04-16; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Direct Oral Anticoagulants (DOACs)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LED+ Haemostatic sponge (Experimental): The experimental group will receive both LED light application and haemostatic sponge treatment
  Interventions: Other: LED light
- Haemostatic sponge only (No Intervention): The active comparator group will receive only the haemostatic sponge

INTERVENTIONS:
Other: LED light — (Dental Light Cure), LED light at wavelengths of 420-480nm and will be applied for 30 seconds at a distance of 1cm from the extraction site
  Arms: LED+ Haemostatic sponge

SUMMARY:
The DENT-DOAC trial is a single-blinded RCT investigating the effectiveness of LED application following dental extractions in patients taking direct oral anticoagulants (DOACs) . The study aims to address a significant clinical challenge, as bleeding following dental extraction is a well-recognized complication in patients taking anticoagulants, and the number of patients taking DOACs requiring dental procedures has increased substantially in recent years.

The trial will be conducted at the Eastman Dental Hospital (EDH-UCLH) and will recruit 50 participants who will be randomly divided into two groups of 25 each. The test group will receive both LED light application and haemostatic sponge treatment, while the control group will receive only the haemostatic sponge.

The study population will include patients taking DOACs (rivaroxaban, apixaban, edoxaban, or dabigatran) and are scheduled for dental extraction. Exclusion criteria include patients using concomitant antithrombotic drugs, those with known allergy to tranexamic acid, pregnant or breastfeeding females, and those recently involved in other research studies. The trial's primary objective is to assess bleeding outcomes in these patients, with secondary objectives including evaluation of bleeding events (early/delayed; minor/moderate/severe) and analysis of associations between bleeding complications and various factors such as type of DOACs, surgical factors, and patient demographics.

The statistical design has been carefully calculated to achieve 90% power to detect both a 50% difference in bleeding events and a 142-second difference in mean bleeding time between groups, with considerations made for a 10% drop-out rate. Patient follow-up will include immediate post-procedure assessment and telephone assessments on days 2 and 7 following the extraction.

ELIGIBILITY:
Inclusion Criteria:

* Taking DOACs (rivaroxaban, apixaban, edoxaban, or dabigatran)
* Listed for dental extraction at EDH
* Willing and able to provide consent

Exclusion Criteria:

* Using concomitant antithrombotic drugs
* Known allergy to tranexamic acid
* Pregnant or breastfeeding females
* Recent involvement in other research studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding time | (Performed intraoperatively) Immediately after intervention (LED) or control (Local Haemostatic Measures) application until bleeding control is achieved (up to 30 minutes)
  Time to achieve bleeding control, measured in seconds or minutes, starting from the application of intervention (LED light) or control (standard local measures) until complete cession of visible bleeding at the site. Timing is recorded by a stopwatch
Number of bleeding events | From the application of intervention (LED) or control up to 7 days post-operatively
  number of bleeding events

CONTACTS AND LOCATIONS:
Locations (1):
- UCL, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/dent-doac/